CLINICAL TRIAL: NCT00728481
Title: The Role Of Gastroesophageal Reflux Disease (GERD) in Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Amy Foxx-Orenstein, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-006685
Record Dates: First submitted 2008-07-15; First posted 2008-08-05 (Estimated); Results first posted 2012-12-06 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Eosinophilic Esophagitis; Gastroesophageal Reflux Disease; EE; GERD
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux | interventions — Esomeprazole; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esomeprazole (Active Comparator): Proton pump inhibitor; Nexium 40mg capsule taken twice daily by mouth for 6 weeks for subjects with positive 24 hour pH study (GERD)
  Interventions: Drug: Esomeprazole
- Budesonide (Active Comparator): Corticosteroid therapy; oral viscous Pulmicort Respules 1 gram taken by mouth orally twice daily (mixed with 1 gram packet of Sucralose [Splenda-registered trademark]) for 6 weeks in subjects with negative 24 hour pH studies (without GERD)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor; Nexium 40mg capsule taken twice daily by mouth for 6 weeks
  Other Names: Nexium
  Arms: Esomeprazole
Drug: Budesonide — Corticosteroid therapy; oral viscous Pulmicort Respules 1 gram taken by mouth orally twice daily (mixed with 1 gram packet of Sucralose [Splenda-registered trademark]) for 6 weeks in subjects with negative 24 hour pH studies (without GERD)
  Other Names: Pulmicort
  Arms: Budesonide

SUMMARY:
The primary aim of this study was to determine the proportion of patients with esophageal eosinophilic infiltration that have objective (measurable) evidence of gastroesophageal reflux disease (GERD).

This study was also done to see if patients that have eosinophilic esophagitis (EE) and GERD would receive relief from taking the medication Nexium or a steroid called Pulmicort.

The study also evaluated the accuracy of pH monitoring (acid exposure) within the esophagus as a predictor of endoscopic, histological and symptomatic response in patients with EE.

DETAILED DESCRIPTION:
Hypotheses:

1. There is a subset of patients with the diagnosis of EE who also have GERD.
2. Patients with both EE and GERD will respond symptomatically and histologically to aggressive gastric acid suppression with a proton pump inhibitor as monotherapy.
3. Swallowed budesonide suspension is effective in treating patients with EE who do not have evidence of GERD.

Participants were randomized based on results of a 24 hour pH study, which determined the average percent time the distal esophagus was exposed to a pH of less than than 4. Subjects with a positive pH result were randomized to esomeprazole or randomized to budesonide, if there was a negative pH result. Studies were interpreted by a single gastroenterologist experienced in reading esophageal pH studies. The percent time the pH monitor detected a pH less than 4 was recorded and an esophageal pH of less than 4 for 4% or greater of the study time was considered abnormal. Note: pH is a measure of acidity or alkalinity (lower numbers are more acid, higher numbers are more alkaline).

Those subjects with GERD (positive pH result) received gastric acid-suppressing medication (esomeprazole 40 mg, twice daily) for 6 weeks. Subjects who did not have GERD (negative pH result) were treated with a corticosteroid designed to coat the esophagus (budesonide suspension 1 mg twice daily) for six weeks. Response to treatment was assessed by esophageal histology and symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 18-80.
2. Patients who carry the diagnosis of Eosinophilic Esophagitis (EE) based on esophageal biopsies obtained within 18 months prior to enrollment with greater than 15 eosinophils (eos) per high power field (hpf) (400 X magnification).
3. Patients who have moderate, severe, or very severe problems swallowing.

Exclusion Criteria:

1. Patients who are currently being treated for EE.
2. Patients who have used topical or systemic corticosteroid therapy for any reason over the past 4 weeks.
3. Patients who have been treated with acid-suppressing medications (Proton Pump Inhibitor or H2 receptor antagonists) within 4 weeks prior to enrollment.
4. Patients with known allergies or hypersensitivity to proton-pump inhibitors or corticosteroids.
5. Patients who have contraindications to the procurement of biopsies including patients how have known bleeding disorders, a history of bleeding diathesis, or who are currently using warfarin or clopidogrel.
6. Patients who have a contraindication to the performance of an esophagogastroduodenoscopy (EGD) including previous cardiopulmonary arrest during an endoscopic procedure.
7. Patients who have contraindications to the performance of ambulatory impedance 24-hour pH testing including patients with oropharyngeal abnormalities that would prohibit the safe passage of the transnasal catheter and patients who are currently using warfarin, have a history of bleeding disorders or bleeding diatheses.
8. Patients who are pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Foxx-Orenstein, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Francis DL, Foxx-Orenstein A, Arora AS, Smyrk TC, Jensen K, Nord SL, Alexander JA, Romero Y, Katzka DA. Results of ambulatory pH monitoring do not reliably predict response to therapy in patients with eosinophilic oesophagitis. Aliment Pharmacol Ther. 2012 Jan;35(2):300-7. doi: 10.1111/j.1365-2036.2011.04922.x. Epub 2011 Nov 24. PMID 22111863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a clinical diagnosis of Eosinophilic Esophagitis (EE) were recruited by mail using a Mayo Clinic proprietary database and also by direct contact in the Mayo Clinic Esophageal Diseases speciality clinic in Rochester, MN. Subjects were enrolled from 3/2009 to 8/2010.
Pre-assignment Details: Patients with esophageal eosinophilic infiltration of greater than or equal to 15 eos/hpf as determined by 4 biopsies of the esophagus, then underwent a 24-hour transnasal catheter-based ambulatory pH study to determine amount of distal esophageal acid exposure, and were placed in one of 2 treatment arms based on positive or negative pH results.
Groups:
- Esomeprazole: Proton pump inhibitor; Nexium 40mg capsule taken twice daily by mouth for 6 weeks for subjects with positive 24 hour pH study
Period: Overall Study
Arm/Group | Esomeprazole | Budesonide
Started | 19 | 32
Completed | 18 | 28
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Study medication non-compliance | 0 | 2
Not completed — Incorrectly assigned to opposite arm | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Budesonide | Total
Number analyzed (Participants) | 19 | 32 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (14.9) | 33.7 (10.4) | 39 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 12 | 19 | 31
Region of Enrollment [Number; unit: participants]
  United States | 19 | 32 | 51
Mean number of eosinophils per high powered field in esophagus [Mean (Standard Deviation); unit: eos/hpf] — Mean eosinophilic density per high power field [eos/hpf] (at 400 x magnification) of four esophageal biopsies each taken from the proximal & distal esophagus at some point 18 months or less prior to study enrollment.
  eos/hpf | 35.6 (24.7) | 46.7 (26.5) | 41.2 (27.7)
Endoscopic evidence of GERD [Number; unit: Participants] — Participants could have had more than one symptom of GERD, or no symptoms of GERD.
  Participants
    Multiple rings (felinization or corrugations) | 14 | 18 | 32
    Hiatal hernia | 15 | 10 | 25
    Erosive esophagitis | 7 | 2 | 9
Number of participants with frequent GERD/dysphagia symptoms [Number; unit: participants] — The GERD portion of the Mayo Dysphagia Questionnaire-30 day (MDQ-30) was used to evaluate the frequency of GERD symptoms. The Mayo Dysphagia Questionnaire is a validated 28 item instrument; 0 = no dysphagia, higher levels indicate greater dysphagia severity.
  Note: 18 of the 19 participants with GERD completed the questionnaire.
  participants
    Frequent symptoms | 15 | 0 | 15
    No or infrequent symptoms | 3 | 17 | 20
    No symptoms | 0 | 15 | 15

OUTCOME MEASURES:

1. Primary Outcome: Histological Response to Treatment
Description: Subjects with Esophageal eosinophilia experiencing a histological response to treatment. Subjects were considered to have histological response to treatment if both sets of biopsies (from the distal and mid-esophagus) had, on average, less than 5 eosinophils per high power field (eos/hpf) at the 6-month biopsies.
Time Frame: Baseline, 6 months
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Budesonide
Number analyzed (Participants) | 18 | 28
Participants
  Subjects with histological response | 11 | 16
  Subjects with nonsignificant histological response | 7 | 12
Statistical Analysis 1: Comparison: Esomeprazole vs Budesonide; Comparison between arms for a histologic response; Test type: Superiority or Other; p = 1.00, Fisher Exact

2. Secondary Outcome: Change in Dysphagia Symptoms in Subjects With Histological Response to Treatment
Description: Dysphagia symptoms were determined based on the Mayo Dysphagia Questionnaire-30 days (MDQ-30), using the question: 'How would you rate the severity of your trouble swallowing in the past 30 days' with a 5 point scale ranging from 'does not bother me at all' to 'very severe, markedly affects my lifestyle'. Symptomatic improvement was defined as only an improvement of 2 levels on this question.
Time Frame: Baseline, 6 months
Population: The analysis population includes only subjects with a histologic response. Subjects were considered to have a histological response to treatment if both sets of biopsies (from distal & mid-esophagus) had, on average, less than 5 eos/hpf.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Budesonide
Number analyzed (Participants) | 11 | 16
Participants
  Dysphagia symptoms improved | 5 | 11
  Dysphagia symptoms did not improve | 6 | 5

3. Secondary Outcome: Change in Dysphagia Symptoms in Subjects With Non-significant Histological Response to Treatment
Description: Dysphagia symptoms were determined based on the Mayo Dysphagia Questionnaire-30 days (MDQ-30), using the question: 'How would you rate the severity of your trouble swallowing in the past 30 days' with a 5 point scale ranging from 'does not bother me at all' to 'very severe, markedly affects my lifestyle'. Patients must have marked a score of 3 or higher corresponding to 'Moderate, cannot be ignored, but does not affect my lifestyle' to be included in the study.
Time Frame: Baseline, 6 months
Population: The analysis population for this item only included subjects with a non-significant histologic response. Subjects were considered to have a histological response to treatment if both sets of 6-month biopsies (from distal & mid-esophagus) had, on average, less than 5 eos/hpf.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Budesonide
Number analyzed (Participants) | 7 | 12
Participants
  Dysphagia symptoms responded to treatment | 6 | 4
  Dysphagia symptoms did not respond | 1 | 8

4. Secondary Outcome: Participants With Presence of Esophageal Rings/Furrows at Six Month Endoscopy
Description: Multiple concentric rings or furrows of the esophagus is an endoscopic finding traditionally ascribed to eosinophilic esophagitis.
Time Frame: Baseline, 6 months
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Budesonide
Number analyzed (Participants) | 18 | 28
participants | 11 | 17

5. Secondary Outcome: Participants With Presence of Erosive Esophagitis at Six Month Endoscopy
Time Frame: Baseline, 6 months
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Budesonide
Number analyzed (Participants) | 18 | 28
participants | 1 | 8

6. Primary Outcome: Symptomatic Response to Treatment
Description: Subjects with Esophageal eosinophilia experiencing a response in their dysphagia symptoms to treatment. Symptomatic improvement in symptoms was defined as a score of at least two levels lower than the baseline dysphagia symptom question on the Mayo Dysphagia Questionnaire-30 days (MDQ-30).
  Dysphagia symptoms were determined based on the MDQ-30 question: 'How would you rate the severity of your trouble swallowing in the past 30 days' with a 5 point scale ranging from 'does not bother me at all' to 'very severe, markedly affects my lifestyle'. Patients must have marked a score of 3 or higher corresponding to 'Moderate, cannot be ignored, but does not affect my lifestyle' to be included in the study.
Time Frame: Baseline, 6 months
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Budesonide
Number analyzed (Participants) | 18 | 28
Participants
  Subjects with response in dysphagia symptoms | 11 | 15
  Subjects with no response in dysphagia symptoms | 7 | 13
Statistical Analysis 1: Comparison: Esomeprazole vs Budesonide; Comparison between arms for a symptomatic response; Test type: Superiority or Other; p = 0.76, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | Esomeprazole | Budesonide
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/28
Other Adverse Events (participants affected / at risk) | 1/18 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esomeprazole (N=18) | Budesonide (N=28)
Hives (Immune system disorders) | 1 (1) | 1 (1) — Subject experienced hives with the initiation of budesonide dosing and withdrew from the study.

LIMITATIONS AND CAVEATS:
The index endoscopy was obtained solely for clinical reasons and could have been done as long as 18 months prior to study enrollment.

A single question on the dysphagia questionnaire was used to assess dysphagia symptom response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No